CLINICAL TRIAL: NCT02161328
Title: EIT: Changes of Pulmonary Ventilation Before and After Tracheotomy
Brief Title: Electric Impedance Tomography Before and After Dilatative Tracheotomy
Status: Completed | Type: Observational
Sponsor: Stefan Kluge (Other)
Responsible Party: Sponsor-Investigator, Stefan Kluge, medical director, Universitätsklinikum Hamburg-Eppendorf
Organization: Universitätsklinikum Hamburg-Eppendorf (Other)
Other Study IDs: EIT2014
Record Dates: First submitted 2014-01-13; First posted 2014-06-11 (Estimated); Last update posted 2020-11-16 (Actual); Status verified 2020-11

CONDITIONS: ICU Patients; Tracheotomy Required

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- ICU patients undergoing a dilatative tracheotomy.
  Interventions: Other: EIT belt

INTERVENTIONS:
Other: EIT belt

SUMMARY:
The changes of local pulmonary ventilation should be registered with an electric impedance tomography (EIT) before and after a dilatative tracheotomy. The hypothesis is that the EIT cannot show changes in local ventilation due to the tracheotomy.

ELIGIBILITY:
Inclusion Criteria:

* treatment on ICU
* indication for tracheotomy
* age between 18 and 85 years
* written to consent

Exclusion Criteria:

* severe chronic pulmonary disease
* cardio pulmonary unstable situation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU patients undergoing an elective dilatative tracheotomy. Before and after tracheotomy the results of EIT will be compared.
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2014-02; Primary Completion 2014-12 (Actual); Study Completion 2015-07-15 (Actual)

PRIMARY OUTCOMES:
volume of ventilation, regional compliance. | Change from Baseline (2 Minutes preoperative) until 2 Minutes postoperative
  measurement starts twenty minutes before surgery and ends after realised recruitment after tracheotomy.

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Universitätsklikum Hamburg Eppendorf, Hamburg
  - Universitätsklinikum Hamburg Eppendorf, Hamburg

REFERENCES:
- [Result] Eichler L, Mueller J, Grensemann J, Frerichs I, Zollner C, Kluge S. Lung aeration and ventilation after percutaneous tracheotomy measured by electrical impedance tomography in non-hypoxemic critically ill patients: a prospective observational study. Ann Intensive Care. 2018 Nov 15;8(1):110. doi: 10.1186/s13613-018-0454-y. PMID 30443867